CLINICAL TRIAL: NCT04730544
Title: Analysis of the Efficacy and Safety of Two Combination Treatment Regimens of Nivolumab and Ipilimumab in Patients With dMMR and / or MSI Metastatic Colorectal Cancer: A GERCOR Open-label, Randomized, Non-comparative, Two-stage Phase II Trial (NIPISAFE).
Brief Title: Two Combination Treatment Regimens of Nivolumab and Ipilimumab in Patients With dMMR and / or MSI mCRC.
Acronym: NIPISAFE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIPISAFE G-106
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Metastatic; MSI-H Colorectal Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm A (Experimental): Treatment for 108 weeks (one cycle = 12 weeks; 9 cycles):
  Nivolumab 480 mg every 4 weeks (27 infusions) and ipilimumab 1 mg/kg every 6 weeks (18 infusions) for a total of 24 months of treatment (or less in case of RECIST progression (PD) or limiting toxicity, whichever occurs first).
  Interventions: Drug: Nivolumab 480mg + Ipilimumab
- Control Arm B (Active Comparator): Induction of 12 weeks (one cycle = 3 weeks; 4 cycles):
  Nivolumab 240 mg and ipilimumab 1 mg/kg every 3 weeks for 4 dosing cycles (4 infusions of nivolumab and ipilimumab), Maintenance of 96 weeks (one cycle = 4 weeks; 24 cycles): Nivolumab 480 mg every 4 weeks for 24 dosing cycles (24 infusions) for a total of 24 months of treatment (or less in case of RECIST progression (PD) or limiting toxicity, whichever occurs first).
  Interventions: Drug: Nivolumab 240 mg + Ipilimumab

INTERVENTIONS:
Drug: Nivolumab 480mg + Ipilimumab — Nivolumab 480 mg q4w + Ipilimumab 1 mg/kg q6w
  Other Names: Opdivo; Yervoy
  Arms: Experimental Arm A
Drug: Nivolumab 240 mg + Ipilimumab — induction phase : Nivolumab 240 mg q3w + Ipilimumab 1 mg/kg q3w and then maintenance : Nivolumab 480 mg q4w
  Other Names: Opdivo
  Arms: Control Arm B

SUMMARY:
NIPISAFE is open-label, phase II study to identify a combination scheme of nivolumab and ipilimumab with a high level of clinical activity, but with a lower toxicity in MSI/dMMR metastatic colorectal cancer patients.

DETAILED DESCRIPTION:
This is a randomized non-comparative two-stage phase II study with a co-primary endpoint (toxicity and progression-free survival) to evaluate two different schemes of the nivolumab and ipilimumab combination in terms of the toxicity and efficacy in MSI/dMMR metastatic colorectal cancer patients in order to identify a combination scheme with a higher level of clinical activity and a lower toxicity.

Patients will be randomized in a 2:1 ratio to receive one of the following treatments:

Experimental ARM A: Nivolumab 480 mg every 4 weeks and ipilimumab 1 mg/kg every 6 weeks for a total of 24 months of treatment Control ARM B: Nivolumab 240 mg and ipilimumab 1 mg/kg every 3 weeks for 4 dosing cycles.

Maintenance of 96 weeks: Nivolumab 480 mg every 4 weeks for 24 dosing cycles for a total of 24 months of treatment (or less in case of RECIST PD or limiting toxicity, whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated patient informed consent form and willingness to comply with all study procedures and availability for the study duration,
2. Age ≥ 18 years,
3. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0, 1, or 2,
4. Histologically or cytologically confirmed colorectal adenocarcinoma,
5. Documented advanced or metastatic disease not suitable for complete surgical resection,
6. At least one measurable lesion as assessed by CT-scan or magnetic resonance imaging (MRI) according to RECIST v1.1 and feasibility of repeated radiological assessments. Participants with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enroll provided the lesion(s) have demonstrated clear progression and can be measured accurately,
7. Deficient mismatch repair (dMMR) and/or Microsatellite instability (MSI) tumor status defined by:

   * Loss of MMR protein expression using immunohistochemistry with four (anti-MLH1, anti-MSH2, anti-MSH6, and anti-PMS2) antibodies Nota Bene (NB): if loss of only one protein, necessary to have Polymerase Chain Reaction (PCR)
   * and/or ≥ two instable markers by pentaplex polymerase chain reaction (BAT-25, BAT-26, NR-21, NR-24, and NR-27), NB: if two instable markers in the pentaplex panel, it is required to present confirmation of the dMMR status by immunohistochemistry or a comparison of the tumor PCR test with matched normal tissue.

   NB: Agreement of the Sponsor (GERCOR) is mandatory to include the patient (the patient's file will be verified to confirm MSI/dMMR status before inclusion [an anonymized fax] and confirmation of a patient's allocation will be sent by mail to the Investigator within 24h),
8. No or one prior line of systemic treatment for metastatic disease:

   * No prior systemic treatment; if patient received neoadjuvant/adjuvant therapy this therapy should be completed > 6 months prior the diagnosis of metastatic or recurrent disease is made,
   * Maximum one prior line of systemic treatment; if patient received one prior line of systemic therapy in the metastatic setting and experienced progression or patient received neoadjuvant/adjuvant therapy and experienced recurrence within ≤ 6 months after completion of therapy,
9. Availability of a representative tumor specimen for exploratory translational research; tumor tissue specimens, either formalin-fixed, paraffin-embedded (FFPE) tissue block or unstained tumor tissue sections (minimum of 30 positively charged slides) from primary or metastatic site must be submitted to the central laboratory,
10. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

    - Hematological status: White blood cell > 2000/µL; Neutrophils > 1500/µL; Platelets > 100.000/µL; Hemoglobin > 9.0 g/dL;

    - Adequate renal function: Serum creatinine level < 150 µM;

    - Adequate liver function: Serum bilirubin ≤ 1.5 x upper normal limit (ULN); Alkaline phosphatase (ALP) ≤ 3 x ULN; Alanine aminotransferase (ALT) ≤ 3.0 x ULN ; Aspartame aminotransferase (AST) ≤ 3.0 x ULN; Prothrombin time (PT)/International normalized ratio (INR) and partial PT (PTT) ≤ 1.5 x ULN unless participants are receiving anticoagulant therapy and their INR is stable and within the recommended range for the desired level of anticoagulation,
11. Females of childbearing potential must have negative serum pregnancy test within 7 days before starting study treatment,
12. Women of childbearing potential should use effective contraception during treatment and 5 months thereafter. Males should use condoms during treatment and 7 months thereafter,
13. Registration in a national health care system ( "Protection Universelle Maladie" (PUMa) included).

Exclusion Criteria:

1. Known brain metastases or leptomeningeal metastases,
2. Persistence of toxicities related to prior chemotherapies grade > 1 (NCI CTCAE v5.0; except alopecia, fatigue, or peripheral sensory neuropathy, which can be grade 2),
3. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, radiotherapy, immunotherapy),
4. Major surgical procedure within 4 weeks prior to initiation of study treatment,
5. Prior treatment with an anti-PD1, anti-programmed death (PD)-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte-associated (CTLA)-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including prior therapy with anti-tumor vaccines or other immuno-stimulatory antitumor agents,
6. Patients receiving any investigational drug, biological, immunological therapy within the previous 28 days before study treatment,
7. Impossibility of submitting to the medical follow-up of the study for geographical, social or psychic reasons,
8. Patients with an active, known or suspected autoimmune disease. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to be enrolled,
9. History of interstitial lung disease or pneumonitis,
10. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease,
11. Prior malignancy active within the previous 3 years, except for:

    * Locally curable cancers that have been apparently cured (e.g. squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast);
    * Lynch syndrome-related non-colorectal cancer in complete remission for > 1 year;
12. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test prior to randomization) virus (HBV) or hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection. Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid.
13. Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
14. Any serious or uncontrolled medical disorder that, in the opinion of Investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the participant to receive protocol therapy, or interfere with the interpretation of study results,
15. Known allergy/hypersensitivity to any component of study agents,
16. Administration of a (attenuated) live vaccine within 28 days of planned start of study therapy of known need for this vaccine during treatment,
17. Patient on tutelage or guardianship or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events grade 3 or 4 at week 24 for two combination schemes. | At week 24
  According to NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Progression-free survival (PFS) at week 24 for two combination schemes. | At week 24 for two combination schemes
  PFS is defined as time from inclusion to the first documented PD determined by the Investigator assessment in accordance to RECIST v1.1 or death due to any cause, whichever occurs first. Alive patients without progression will be censored at the last tumor assessment, either during study treatment period or during follow-up period.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | Assessed up to 80 months
  All grade and severe toxicities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Overall response rate (ORR) | At weeks 24 and 48, and at 2 years
  To assess ORR of two combination schemes (RECIST v1.1),
PFS of two combination schemes according to RECIST v1.1 | At week 48 and at 2 years
  PFS is defined as time from inclusion to the first documented PD determined by the Investigator assessment in accordance to RECIST v1.1 or death due to any cause, whichever occurs first. Alive patients without progression will be censored at the last tumor assessment, either during study treatment period or during follow-up period.
PFS of two combination schemes according to Immune Response Evaluation Criteria In Solid Tumors (iRECIST) | At weeks 24 and 48, and at 2 years
  PFS is defined as time from inclusion to the first documented PD determined by the Investigator assessment in accordance to RECIST v1.1 or death due to any cause, whichever occurs first. Alive patients without progression will be censored at the last tumor assessment, either during study treatment period or during follow-up period.
Overall survival (OS) of two combination schemes (RECIST v1.1), | At week 48 and at 2 years
  OS is defined as the time between inclusion and death.
Percentage of patients who received immune modulating concomitant medication | Until the study treatment end - 48 months
  To evaluate the percentage of patients who received immune modulating concomitant medication (e.g., corticosteroids, infliximab, mycophenolate mofetil).
Percentage of patients who received hormonal replacement therapy for immune-related endocrine toxicities | Until the study treatment end - 48 months
  To evaluate the percentage of patients who received hormonal replacement therapy for immune-related endocrine toxicities.
Median time to onset, median time to resolution (grade 3-4) of serious adverse event (SAEs) and Treatment-related adverse events (TRAEs), | Up to 80 months
  To assess median time to onset and median time to resolution of serious AEs (SAEs) and TRAEs (grade 3-4).
Time to Health-related quality of life (HRQoL) score definitive deterioration (TUDD) | assessed up 48 months
  TUDD is defined as the time interval between randomization and the first occurrence of a decrease in quality of life questionnaire (QLQ)-C30 score ⩾5 points without any further improvement in Quality of life (QoL) score ⩾5 points or any further available QoL data. TUDD will be estimated using the Kaplan-Meier method and the long-rank test. Cox regression analyses will be used to identify HRQoL items influencing TUDD. All analyses will be done on the HRQoL population.

CONTACTS AND LOCATIONS:
Overall Officials: Romain COHEN, MD, Principal Investigator — Saint Antoine Hospital
Locations (19):
- France (19):
  - Institut Sainte Catherine, Avignon
  - CHU Jean Minjoz, Besançon
  - CHU Morvan, Brest
  - Hôpital Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - Clinique Victor Hugo-Centre jean Bernard, Le Mans
  - Hopital Franco-Britannique - Fondation Cognacq-Jay, Levallois-Perret
  - CHRU Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital de la Timone, Marseille
  - ICM Val d'Aurelle, Montpellier
  - CHU Nantes- Hôtel Dieu, Nantes
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Bordeaux - Hôpital Haut Lévêque, Pessac
  - CHU Poitiers, Poitiers
  - Hôpital Robert Debré, Reims
  - CHU Toulouse - IUCT Rangueil -Larrey, Toulouse

IPD SHARING:
Plan to Share IPD: No